CLINICAL TRIAL: NCT00363857
Title: A 12-Week, Double-Blind, Placebo Controlled, Parallel Group Study to Assess the Efficacy and Safety of Ropinirole in Patients Suffering From Restless Legs Syndrome (RLS)
Brief Title: A Clinical Research Study Testing Ropinirole Treatment for Restless Legs Syndrome
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 101468/249
Record Dates: First submitted 2006-08-11; First posted 2006-08-15 (Estimated); Last update posted 2016-10-17 (Estimated); Status verified 2016-10

CONDITIONS: Restless Legs Syndrome (RLS); Restless Legs Syndrome
Keywords: fatigue; sleep; sleep disorder; Legs; RLS; Restless Legs Syndrome; Ropinirole
MeSH Terms: conditions — Restless Legs Syndrome; Fatigue; Sleep Wake Disorders | interventions — ropinirole

INTERVENTIONS:
Drug: Ropinirole

SUMMARY:
A 14-Week clinical research study to compare the effectiveness and safety of ropinirole and placebo (an inactive sugar pill) in the treatment of patients with Restless Legs Syndrome (RLS) in the United States.

ELIGIBILITY:
Inclusion criteria:

* Patients diagnosed with Restless Legs Syndrome (RLS) with symptoms such as: uncomfortable or "creepy-crawly" sensations in your legs, overwhelming urge to move your legs to relieve these sensations, sensations go away when you move your legs, or trouble falling asleep or staying asleep because of these symptoms.
* Patients must give written informed consent prior to any specific study procedures.

Exclusion criteria:

* Patients who suffer from narcolepsy, sleep terror disorder, sleepwalking disorder, or a breathing related sleep disorder.
* Patients diagnosed with renal failure (end-stage renal disease) iron deficient anemia or pregnancy.
* Patients suffering from other movement disorders (i.e. Parkinson's Disease).
* Patients who have medical conditions such as diabetes, peripheral neuropathy, rheumatoid arthritis, or fibromyalgia syndrome.
* Participation in any clinical drug or device trial in the last three months.

Other inclusion or exclusion criteria to be evaluated by the physician.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Actual)
Dates: Start 2003-08; Primary Completion 2004-05 (Actual); Study Completion 2004-05 (Actual)

PRIMARY OUTCOMES:
Improvement in RLS severity rating scale at Week 12

SECONDARY OUTCOMES:
Percentage of patients who were much improved or very much improved on an overall clinical rating scale at Week 12.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (47):
- United States (47):
  - GSK Investigational Site, Alabaster, Alabama
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Jasper, Alabama
  - GSK Investigational Site, Tuscaloosa, Alabama
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Little Rock, Arkansas
  - GSK Investigational Site, Berkeley, California
  - GSK Investigational Site, La Jolla, California
  - GSK Investigational Site, Northridge, California
  - GSK Investigational Site, Oxnard, California
  - GSK Investigational Site, Redondo Beach, California
  - GSK Investigational Site, Santa Monica, California
  - GSK Investigational Site, Stanford, California
  - GSK Investigational Site, Aurora, Colorado
  - GSK Investigational Site, Danbury, Connecticut
  - GSK Investigational Site, Boca Raton, Florida
  - GSK Investigational Site, Largo, Florida
  - GSK Investigational Site, Pembroke Pines, Florida
  - GSK Investigational Site, St. Petersburg, Florida
  - GSK Investigational Site, Tampa, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Augusta, Georgia
  - GSK Investigational Site, Macon, Georgia
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Elk Grove Village, Illinois
  - GSK Investigational Site, Louisville, Kentucky
  - GSK Investigational Site, Southfield, Michigan
  - GSK Investigational Site, Henderson, Nevada
  - GSK Investigational Site, Lebanon, New Hampshire
  - GSK Investigational Site, Albuquerque, New Mexico
  - GSK Investigational Site, Schenectady, New York
  - GSK Investigational Site, Raleigh, North Carolina
  - GSK Investigational Site, Columbus, Ohio
  - GSK Investigational Site, Concinnati, Ohio
  - GSK Investigational Site, Dublin, Ohio
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - GSK Investigational Site, Portland, Oregon
  - GSK Investigational Site, Lafayette Hill, Pennsylvania
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Columbia, South Carolina
  - GSK Investigational Site, Nashville, Tennessee
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Plano, Texas
  - GSK Investigational Site, Alexandria, Virginia
  - GSK Investigational Site, Norfolk, Virginia
  - GSK Investigational Site, Walla Walla, Washington

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Informed Consent Form: 101468/249 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 101468/249 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 101468/249 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 101468/249 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 101468/249 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 101468/249 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 101468/249 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register